CLINICAL TRIAL: NCT01331863
Title: Replacement of the Airways and/or the Pulmonary Vessels Using a Cryopreserved Arterial Allograft
Brief Title: Airway and/or Pulmonary Vessels Transplantation
Acronym: TRACHBRONCAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P091203
Record Dates: First submitted 2011-04-07; First posted 2011-04-08 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2017-08

CONDITIONS: Lung Cancer; Tracheal Neoplasm; Tracheal Stenosis
Keywords: Bronchial disease; Lung cancer surgery; Aorta/aortic Allograft; homograft; Tracheal disease; Benign; Malignant
MeSH Terms: conditions — Lung Neoplasms; Tracheal Neoplasms; Tracheal Stenosis; Bronchial Diseases; Tracheal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm surgery (Experimental): Airway and/or pulmonary Vessels Transplantation
  Interventions: Procedure: Airway and/or pulmonary Vessels Transplantation

INTERVENTIONS:
Procedure: Airway and/or pulmonary Vessels Transplantation — Use of a stent-supported aortic allograft to prevent pneumonectomy in lung cancer SURGERY

SUMMARY:
* First study (BRONC-ART) The purpose of this prospective study is to evaluate the 90-day morbidity and mortality rates of bronchial transplantation using cryopreserved aortic allograft in proximal lung cancer surgery. The investigators hypothesize that this stage 1-2 surgical innovation could be safe and effective in order to reduce the 90-day morbidity and mortality rates compared to those observed with pneumonectomy, especially when some factors are present: age > 70 years, right side, neoadjuvant chemoradiotherapy.
* Current study (TRACHEO BRONC-ART) The BRONC-ART study was extended to major (malignant or benign) lesions of the trachea requiring airway transplantation.

For these patients, resection followed by direct end to end anastomosis is not possible or at high risk.

DETAILED DESCRIPTION:
Surgery remains the best option for curative treatment of early stages Non-Small Cell Lung Cancer (NSCLC). Peripheral tumors are usually resected using lobectomy with a low 90-day morbidity and mortality rate (2%). Central NSCLC often require a pneumonectomy with a high 90-day morbidity and mortality rate (up to 24%), especially when some factors are present: age > 70 years, right side, neoadjuvant chemoradiotherapy. On the other hand, bronchoplastic lobectomies have been proposed in order to avoid pneumonectomy. However, more than fifty years after their first description, bronchoplastic lobectomies remain uncommon (<1% of all pulmonary resection). This could be explained by some technical difficulties showing the potential interest of a bronchial substitute. In a 10-year research phase on a sheep model (n=108), we demonstrated that aortic grafts could be valuable substitutes for tracheobronchial replacement. We observed a progressive transformation of the aortic tissue into airway tissue comprising epithelium and regenerated cartilage. The technique was extended to clinical tracheal replacement by us and others with encouraging results. We proposed to evaluate the feasibility of the use of a stent-supported cryopreserved aortic allograft as a bronchial substitute to prevent pneumonectomy and its associated high mortality rate in NSCLC surgery. Primary outcome will be the 90-day mortality. Secondary outcomes will be the postoperative complications, the 90-day morbidity. This prospective open study will include 20 to 30 patients according to eligibility criteria (see below). The operation will consist of the curative resection of the NSCLC followed by the replacement of a bronchial segment using a cryopreserved allograft in order to re-implant a functional pulmonary lobe. A stent will be placed in the graft to prevent airway collapse.

-Current study (TRACHEO BRONC-ART) The BRONC-ART study was extended to major (malignant or benign) lesions of the trachea requiring airway transplantation. For these patients, resection followed by direct end to end anastomosis is not possible or at high risk.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥18 years and patient capable of giving consent to the carrying out of a medical research procedure
* patient with proximal Lung Cancer (LC) requiring surgical resection (carinal resection, pneumonectomy, bronchoplastic lobectomy) after neoadjuvant chemotherapy or not and with adequate preoperative lung function tests
* or patient with proximal LC requiring a pneumonectomy without adequate preoperative lung function tests
* patients with extended lesions malignant or benign of the trachea without bronchitic lesion and who are in therapeutic impasse.
* or patient older than 70 years with proximal LC requiring a pneumonectomy
* decision made by a multidisciplinary team
* patient information and consent

Exclusion Criteria:

* patient age < 18 years or patient not capable of giving consent to the carrying out of a medical research procedure
* patient with proximal or peripheral LC requiring a simple lobectomy
* patient with unresectable LC because of major local involvement, N3 and/or M1 status(with the exception of a unique resectable brain metastasis)
* patient with tracheal lesion that can be isolated from a simple resection anastomosis tracheal
* iodine allergy
* preoperative evaluation not allowing a simple lobectomy
* patient not affiliated to the French Social Security System

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
90-day mortality | 3 months

SECONDARY OUTCOMES:
90-day morbidity | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel MARTINOD, Pr, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris, Hôpital Avicenne, CHU Paris-Seine-Saint-Denis, Bobigny, Seine-Saint-Denis, France

REFERENCES:
- [Derived] Martinod E, Chouahnia K, Radu DM, Joudiou P, Uzunhan Y, Bensidhoum M, Santos Portela AM, Guiraudet P, Peretti M, Destable MD, Solis A, Benachi S, Fialaire-Legendre A, Rouard H, Collon T, Piquet J, Leroy S, Venissac N, Santini J, Tresallet C, Dutau H, Sebbane G, Cohen Y, Beloucif S, d'Audiffret AC, Petite H, Valeyre D, Carpentier A, Vicaut E. Feasibility of Bioengineered Tracheal and Bronchial Reconstruction Using Stented Aortic Matrices. JAMA. 2018 Jun 5;319(21):2212-2222. doi: 10.1001/jama.2018.4653. PMID 29800033